CLINICAL TRIAL: NCT04700267
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Orally Administered GLPG3970 for 12 Weeks in Adult Subjects With Active Systemic Lupus Erythematosus
Brief Title: A Study Evaluating the Effects of GLPG3970 Given as Oral Treatment for 12 Weeks in Adults With Systemic Lupus Erythematosus
Acronym: TAPINOMA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped on business grounds
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG3970-CL-102; 2020-001820-32 (EudraCT Number)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG3970 (Experimental): One dose level of GLPG3970
  Interventions: Drug: GLPG3970 film-coated tablet
- Placebo (Placebo Comparator): One dose level of Placebo
  Interventions: Drug: Placebo film-coated tablet

INTERVENTIONS:
Drug: GLPG3970 film-coated tablet — GLPG3970 for oral administration
  Arms: GLPG3970
Drug: Placebo film-coated tablet — Placebo for oral administration
  Arms: Placebo

SUMMARY:
This is a first exploration of GLPG3970 in subjects with active systemic lupus erythematosus (SLE) to evaluate the effect on disease biomarkers and to determine its pharmacokinetics (PK) profile, safety and tolerability, and pharmacodynamics (PD) biomarkers related to the investigational product (IP) mechanism of action and the pathophysiology of SLE.

ELIGIBILITY:
Inclusion Criteria:

* SLE diagnosis defined by American College of Rheumatology (ACR) 1997 criteria ≥4
* Active arthritis in >=4 active joints (according to 28 joint count) and/or cutaneous lupus erythematosus disease area and severity index (CLASI) score >=6.
* Anti-dsDNA antibodies >15 IU/mL.
* Stable standard-of-care (SoC) therapy (defined as no change in prescription for at least 2 weeks prior to first IP dosing) consisting of the following permitted SoC medications:

  * Corticosteroids <=20 mg/day (prednisone or equivalent) for at least 2 weeks prior to first IP dosing; AND/OR
  * Non-steroidal anti-inflammatory drug (NSAIDs); AND/OR
  * One single antimalarial at a stable dose (hydroxychloroquine <=5 mg/ kg/day, quinacrine 100 mg/day, or chloroquine 2.3 mg/kg/day) for at least 8 weeks prior to first IP dosing; AND/OR
  * One single immunosuppressant at a stable dose (azathioprine (AZA) <=2 mg/kg/day, methotrexate (MTX) <=20 mg/week, or mycophenolate mofetil (MMF) <=2 g/day) for at least 8 weeks prior to first IP dosing.
* estimated glomerular filtration rate (eGFR) >=60 mL/min (according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI))

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Lupus nephritis >= Class III
* Severe organ manifestation or life-threatening lupus disease (active severe central nervous system lupus, severe pleuro-pericarditis, severe vasculitis).
* Severe acute respiratory syndrome coronavirus disease 2 (SARS-CoV-2) infection >0
* Unstable condition not related to SLE
* Systemic inflammatory condition other than SLE such as, but not limited to rheumatoid arthritis (RA), spondyloarthropathy, Crohn's disease, ulcerative colitis, or psoriatic arthritis
* Sjögren's syndrome and/or antiphospholipid antibody syndrome who do not require treatment with any prohibited medication are NOT excluded.
* Active systemic infection
* Poorly controlled chronic cardiac, pulmonary, or renal disease.
* Known or suspected history of or a current immunosuppressive condition, or a history of invasive opportunistic infections
* Treatment with disallowed therapies

This list only contains the key exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers associated with disease anti-dsDNA | Between Day 1 and 104
  To characterize the PD of GLPG3970 compared to placebo in adult subjects with active SLE
Change in biomarkers associated with disease complement component 3 (C3), and complement component 4 (C4) | Between Day 1 and 104
  To characterize the PD of GLPG3970 compared to placebo in adult subjects with active SLE
Number, incidence, and severity of treatment-emergent adverse events (TEAEs) | From screening through study completion, an average of 5 months
  To evaluate the safety and tolerability of GLPG3970 compared to placebo in adult subjects with active SLE

SECONDARY OUTCOMES:
Observed GLPG3970 plasma trough concentrations (Ctrough) | Between Day 1 and 87
  To characterize the PK of GLPG3970 in adult subjects with active SLE

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Vincent, MD, Study Director — Galapagos NV
Locations (14):
- Bulgaria (3):
  - Medical center Medconsult Pleven, Pleven
  - UMHAT-Plovdiv AD, Plovdiv
  - UMHAT Sv. Ivan Rilski EAD, Sofia
- ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- Poland (4):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Medycyna Kliniczna, Warsaw
  - FutureMeds sp. Z o. o., Wroclaw
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- Ukraine (5):
  - Medical Centre of Ltd Liability Comp, Kyiv
  - Multidisciplinary Medical Center of Odesa National Medical University, Odesa
  - N.I.Pirogov Vinnytsia Reg Council, Vinnytsia
  - SRI of Invalid Rehabilitation, Vinnytsia
  - LLC Suchasna klinika, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No